CLINICAL TRIAL: NCT05211492
Title: Acute and Chronic Pain After One-stage Hybrid Arrhythmia Ablation Surgery: A Study on the Presence of Chronic Pain After Hybrid Ablation and Factors That May be Associated
Brief Title: Acute and Chronic Pain After One-stage Hybrid Arrhythmia Ablation Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients were recruited
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pain 1StageHybride Ablation
Record Dates: First submitted 2021-12-22; First posted 2022-01-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2023-04

CONDITIONS: Arrythmia; Chronic Pain; Acute Pain; Post Operative Pain
MeSH Terms: conditions — Arrhythmias, Cardiac; Chronic Pain; Acute Pain; Pain, Postoperative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: There are 3 groups. 1 chronic pain, 2 acute pain, 3 no pain
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chronic pain (Other)
  Interventions: Other: Questionnaire
- Acute pain (Other)
  Interventions: Other: Questionnaire
- Control group (Other)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients are asked to fill in an online questionnaire concerning their postoperative pain.

SUMMARY:
After one-stage hybrid arrhythmia ablation surgery there are possible side effects like acute and chronic pain. There is a lot of research surrounding these pains but not specifically after one-stage hybrid arrhythmia ablation surgery. The investigators want to research factors that may be associated with the absence of chronic pain after hybrid ablation include ketamine, peroperative opioids, loco-regional blocks, neuraxial blocks, wound infiltration, postoperative patient-controlled analgesia. The presence of corticosteroids or NSAIDS, will also be evaluated. Furthermore, non-adaptable factors such as genetics complicate the onset of chronic post-operative pain. Taking existing knowledge in this field into account, incidence risk as well as acute pain duration and intensity and their effects on chronic pain will become the primary focus of this study.

The investigators will contact all patients who had a one-stage hybrid arrhythmia ablation surgery at UZ Brussels. Participants will be sent a questionnaire with a consent form in and a survey asking about their pain 3 months postop and their current pain management therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* he/she must understand and read the Dutch, French or English language
* be able to digitally agree to participate in the study
* had to have a one stage hybrid procedure at least three months ago
* have an ASA score of I, II or III.

Exclusion Criteria:

* Patients with previously known chronic pain syndromes, fibromyalgia, complex regional pain syndrome are excluded.
* Subjects with previous known chronic conditions such as diabetes neuropathy, rheumatoid arthri-tis, … are also excluded.
* Subject are excluded if they underwent a surgical treatment within the observed period.
* Patients are excluded when under treatment with chemotherapy/radiotherapy
* Pregnant patients are also excluded.
* Patients with known psychological conditions such as depression are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with acute pain after one stage hybrid ablation. | 3 months postop
  How many patients have acute pain after surgery
Number of patients with chronic pain after one stage hybrid ablation. | 3 months postop
  How many patients have acute pain after surgery

SECONDARY OUTCOMES:
Intensity of immediate pain following one stage hybrid ablation | 3 days
  How painful on a numeric pain scale rating of 0 to 10 is the immediate pain post operation? 10 being the worst pain ever felt and 0 being totally painfree.
Duration of immediate pain following one stage hybrid ablation | 3 days
  How long does the immediate pain post operation last?
Intensity of acute and chronic pain after receiving an advance anesthesiologic pain block. | 3 months
  How painful on a numeric pain scale rating of 0 to 10 is the acute or chronic pain post operation? 10 being the worst pain ever felt and 0 being totally pain free.
Intensity of acute and chronic pain after administration of ketamine. | 3 months
  How painful on a numeric pain scale rating of 0 to 10 is the acute or chronic pain post operation? 10 being the worst pain ever felt and 0 being totally pain free.
Intensity of acute and chronic pain after treatment with opioids. | 3 months
  How painful on a numeric pain scale rating of 0 to 10 is the acute or chronic pain post operation? 10 being the worst pain ever felt and 0 being totally pain free.
Intensity of acute and chronic pain after placing of a thorax drain post operatively. | 3 months
  How painful on a numeric pain scale rating of 0 to 10 is the acute or chronic pain post operation? 10 being the worst pain ever felt and 0 being totally pain free.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No